CLINICAL TRIAL: NCT02899884
Title: Characterisation and Epidemiology of Breakthrough Cancer Pain in Spain
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: Fentanyl-5001; CARPEDIO Study (Other: Other)
Record Dates: First submitted 2016-09-09; First posted 2016-09-14 (Estimated); Results first posted 2019-11-22 (Actual); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Breakthrough Cancer Pain
Keywords: Drug Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort 1: Participants with cancer pain that is adequately controlled with opioids were observed for a period of 1 month in this observational study.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention

SUMMARY:
The purpose of this study is to determine the prevalence of breakthrough cancer pain and characterize breakthrough cancer pain in an unselected, representative cohort of cancer outpatients with or without pain who attend consultations.

DETAILED DESCRIPTION:
This study has been designed as a non-interventional, non post-authorization, cross-sectional, epidemiological study to determine the prevalence of breakthrough cancer pain and characterize breakthrough cancer pain in an non-selected, representative cohort of cancer outpatients with or without pain.

The study enrolled 3765 patients. This multicenter trial will be conducted in Spain. Data from participants will be collected through questionnaire and medical history in a single visit (up to 1 month).

ELIGIBILITY:
Inclusion Criteria:

* Participants≥ 18 years old
* Participants with baseline cancer pain that is adequately controlled with opioids
* Presence of episodes of breakthrough pain associated with the cancer pain
* Meeting the diagnostic criteria for breakthrough cancer pain (participant history and Portenoy's criteria) and the Davies algorithm
* Participants who are not receiving treatment for breakthrough cancer pain. It is not permitted the inclusion of participants receiving treatment for breakthrough cancer pain in order to avoid bias that may affect the characterization or taxonomy of breakthrough cancer pain
* Signing of the informed consent

Exclusion Criteria:

* Severe mental illness
* Any medical condition or situation complicating the collection of study data as determined by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with cancer pain will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 3765 (Actual)
Dates: Start 2016-11-14 (Actual); Primary Completion 2018-04-04 (Actual); Study Completion 2018-07-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (36):
- Spain (36):
  - Hospital General Universitario de Elda-Virgen de La Salud, Elda, Alicante
  - Hospital Universitario San Juan de Alicante, San Juan, Alicante
  - Hospital Universitari Son Espases, Palma de Mallorca, Balearic Islands
  - Hospital Son Llatzer, Palma de Mallorca, Balearic Islands
  - Hospital Universitari Germans Trias I Pujol de Badalona, Badalona, Barcelona
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital de Especialidades de Puerto Real, Puerto Real, Cadiz
  - Hospital Universitario de Gran Canaria Dr. Negrin, Las Palmas de Gran Canaria, Canary Islands
  - Complejo Hospitalario Universitario Insular-Materno Infantil, Las Palmas de Gran Canarias, Canary Islands
  - Hospital Universitario Nuestra Senora de Candelaria, Santa Cruz de Tenerife, Canary Islands
  - Hospital de Alta Resolucion de Guadix, Guadix, Granada
  - Hospital Universitario Principe de Asturias, Alcalá de Henares, Madrid
  - Hospital Universitario Puerta de Hierro, Majadahonda, Majadahonda, Madrid
  - Hospital Quiron Madrid, Pozuelo de Alarcón, Madrid
  - Complejo Hospital Costa Del Sol, Marbella, Malaga
  - Hospital General Universitario Santa Lucia, Cartagena, Murcia
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - Hospital Los Montalvos, Carrascal de Barregas, Salamanca
  - Complexo Hospitalario Universitario A Coruna, A Coruña
  - Centro Oncoloxico de Galicia, A Coruña
  - Hospital Torrecardenas, Almería
  - Hospital Puerta Del Mar, Cadiz
  - Hospital Reina Sofia, Córdoba
  - Hospital Universitario Virgen de Las Nieves, Granada
  - Complejo Hospitalario de Jaen, Jaén
  - Hospital Universitario de La Princesa, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Complejo Hospitalario Regional de Malaga, Málaga
  - Hospital Virgen de La Victoria, Málaga
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Nuestra Senora de Valme, Seville
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital General Universitario de Valencia, Valencia
  - Hospital Universitario Doctor Peset, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available for all interventional studies after applicable marketing approvals and commercial availability have been received (or program is completely terminated), an opportunity for the primary publication of the research and final report development has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 32 investigative sites in Spain from 14 November 2016 to 16 July 2018.
Pre-assignment Details: Participants with a diagnosis of cancer pain were enrolled and observed to characterize the participants with breakthrough pain.
Period: Overall Study
Arm/Group | Cohort 1
Started | 3765
Completed | 3765
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Arm/Group | Cohort 1
Number analyzed (Participants) | 3765
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Number analyzed is the number of participants with data available for this baseline measure.
  years
    number analyzed (Participants) | 3721
    (all) | 65 (13)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Number analyzed is the number of participants with data available for this baseline measure.
  Participants
    number analyzed (Participants) | 3736
    Female | 1789
    Male | 1947
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Spain | 3765

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Cancer Participants With Breakthrough Cancer Pain From the Total Number of Cancer Participants Seen in Consultation
Description: Breakthrough cancer pain was defined as the temporary exacerbation of pain occurring either spontaneously or in relation to a specific, predictable or unpredictable trigger in spite of relatively stable and adequately controlled baseline pain.
Time Frame: Month 1
Population: Prevalence Study Population included participants with the prevalence of breakthrough cancer pain for whom data was collected in prevalence form in the database.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1
Number analyzed (Participants) | 3765
percentage of participants | 14.3 [13.2 to 15.4]

2. Primary Outcome: Percentage of Cancer Participants With Breakthrough Cancer Pain From the Number of Cancer Participants With Pain Seen in Consultation
Description: as for outcome 1
Time Frame: Month 1
Population: Participants with cancer pain from the Prevalence Study Population, participants with the prevalence of breakthrough cancer pain for whom data was collected in prevalence form in the database.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1
Number analyzed (Participants) | 1117
percentage of participants | 48.3 [45.3 to 51.2]

3. Secondary Outcome: Number of New Participants Diagnosed With Breakthrough Cancer Pain From the Total Number of Cancer Participants Seen in Consultation
Description: Participants diagnosed during the study and were not diagnosed previously were reported as new participants with breakthrough cancer pain. Breakthrough cancer pain was defined as the temporary exacerbation of pain occurring either spontaneously or in relation to a specific, predictable or unpredictable trigger in spite of relatively stable and adequately controlled baseline pain.
Time Frame: Month 1
Population: Prevalence Study Population included participants with the prevalence of breakthrough cancer pain for whom data was collected in prevalence form in the database. Number analyzed is the total number of participants with data available for the time of diagnosis of breakthrough cancer pain.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1
Number analyzed (Participants) | 3765
Participants | 105

4. Secondary Outcome: Percentage of New Participants Diagnosed With Breakthrough Cancer Pain From the Number of Cancer Participants With Pain Seen in Consultation
Description: as for outcome 3
Time Frame: Month 1
Population: Participants with cancer pain from the Prevalence Study Population, participants with the prevalence of breakthrough cancer pain for whom data was collected in prevalence form in the database, with data available for the time of diagnosis of breakthrough cancer pain.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1
Number analyzed (Participants) | 544
percentage of participants | 19.3 [16.0 to 22.6]

5. Secondary Outcome: Pain Characterization With the Alberta Breakthrough Pain Assessment
Description: The Alberta Breakthrough Pain Assessment Tool (ABPAT) consisted of a participant's self-reporting section (15 questions) out of which 4 questions of the tool were not included as they were related to the treatment for breakthrough cancer pain. The questions included: Q1-Relationship to baseline pain, Q2a-Last time experienced, Q3b-Frequency, Q4b-Intensity of pain at peak, Q5-Location (most frequent - ≥5%), Q6-Quality (those present in ≥20%), Q7-Time from onset to peak intensity, Q8-Time from onset [take medication] to end of episode, Q9-Cause(s) (triggers) (Those present in ≥20%), Q10-Predictability, Q11-General relief (those present in ≈20% or more participants) and questions completed by nurse/physician (N/P), Q1-Etiology of breakthrough pain, Q2-Inferred pathophysiology of breakthrough pain. Percentage of participants were categorized into the answers for each of these questions.
Time Frame: Month 1
Population: Participants from Prevalence Study Population, participants with the prevalence of breakthrough cancer pain for whom data was collected in prevalence form in the database with breakthrough cancer pain who did not take any treatment for it and who administered the scale. Number analyzed is the participants with data available for the given question.
Measure: Number; unit: percenatge of participants
Arm/Group | Cohort 1
Number analyzed (Participants) | 195
percenatge of participants
  Q1, Brief Flare-up of Baseline Pain: number analyzed (Participants) | 190
  Q1, Brief Flare-up of Baseline Pain | 53.2
  Q1, Different from Baseline Pain: number analyzed (Participants) | 190
  Q1, Different from Baseline Pain | 36.3
  Q1, Not Sure: number analyzed (Participants) | 190
  Q1, Not Sure | 10.5
  Q2a, Today: number analyzed (Participants) | 194
  Q2a, Today | 57.7
  Q2a, Yesterday: number analyzed (Participants) | 194
  Q2a, Yesterday | 33.0
  Q2a, Before then: number analyzed (Participants) | 194
  Q2a, Before then | 9.3
  Q3b, Usual: number analyzed (Participants) | 182
  Q3b, Usual | 62.6
  Q3b, Better: number analyzed (Participants) | 182
  Q3b, Better | 8.4
  Q3b, Worse: number analyzed (Participants) | 182
  Q3b, Worse | 29.1
  Q4b, Mild: number analyzed (Participants) | 194
  Q4b, Mild | 1.5
  Q4b, Moderate: number analyzed (Participants) | 194
  Q4b, Moderate | 16.0
  Q4b, Severe: number analyzed (Participants) | 194
  Q4b, Severe | 82.5
  Q5, Lumbar | 20.0
  Q5, Hips | 6.7
  Q5, Abdominal | 6.7
  Q5, Back | 6.2
  Q5, Thoracolumbar | 5.1
  Q5, Thoracic | 5.1
  Q6, Stabbing | 57.9
  Q6, Splitting | 29.7
  Q6, Sharp | 29.2
  Q6, Punishing-Cruel | 27.2
  Q6, Heavy | 26.7
  Q6, Hot-Burning | 25.6
  Q6, Fearful | 21.5
  Q7, More than 0 and Up to 10 Minutes | 57.4
  Q7, More than 10 and Up to 30 Minutes | 24.1
  Q7, More than 30 Minutes | 8.2
  Q7, It is Hard to Say Exactly When It Started | 10.3
  Q8, More than 0 and Up to 10 minutes: number analyzed (Participants) | 192
  Q8, More than 0 and Up to 10 minutes | 18.8
  Q8, More than 10 and Up to 30 minutes: number analyzed (Participants) | 192
  Q8, More than 10 and Up to 30 minutes | 37.5
  Q8, More than 30 Minutes: number analyzed (Participants) | 192
  Q8, More than 30 Minutes | 33.3
  Q8, I am Not on Any Breakthrough Pain Medication: number analyzed (Participants) | 192
  Q8, I am Not on Any Breakthrough Pain Medication | 10.4
  Q9, Movement in Bed | 33.3
  Q9, Walking | 31.8
  Q9, Standing | 29.7
  Q9, Sitting | 19.5
  Q9, Coughing | 19.5
  Q10, I Can Never Predict When It will Occur | 19.5
  Q10, I Can Rarely Predict When It will Occur | 17.4
  Q10, I Can Sometimes Predict When It will Occur | 20.5
  Q10, I Can Often Predict When It will Occur | 30.3
  Q10, I Can Always Predict When It will Occur | 12.3
  Q11, Lying | 37.4
  Q11, Use of Scheduled Pain Medication | 19.5
  Q11, Unsure | 19.5
  Q1:N/P,Pain Related to the Site of Active Cancer: number analyzed (Participants) | 186
  Q1:N/P,Pain Related to the Site of Active Cancer | 78.0
  Q1:N/P, Related to Body/Cancer's Systemic Effects: number analyzed (Participants) | 186
  Q1:N/P, Related to Body/Cancer's Systemic Effects | 5.9
  Q1:N/P,Pain Related to Anticancer Treatment: number analyzed (Participants) | 186
  Q1:N/P,Pain Related to Anticancer Treatment | 9.7
  Q1:N/P,Pain Caused by a Concurrent Disorder: number analyzed (Participants) | 186
  Q1:N/P,Pain Caused by a Concurrent Disorder | 4.8
  Q1:N/P,Unknown or Uncertain at this Time: number analyzed (Participants) | 186
  Q1:N/P,Unknown or Uncertain at this Time | 1.6
  Q2:N/P,Somatic Nociceptive: number analyzed (Participants) | 186
  Q2:N/P,Somatic Nociceptive | 55.9
  Q2:N/P,Visceral Nociceptive: number analyzed (Participants) | 186
  Q2:N/P,Visceral Nociceptive | 16.1
  Q2:N/P,Neuropathic: number analyzed (Participants) | 186
  Q2:N/P,Neuropathic | 19.9
  Q2:N/P,Unknown or Uncertain at this Time: number analyzed (Participants) | 186
  Q2:N/P,Unknown or Uncertain at this Time | 8.1

6. Secondary Outcome: Pain Severity and Pain Interference as Assessed by Brief Pain Inventory (BPI) Questionnaire Score
Description: The BPI questionnaire was used to assess the pain intensity (4 items) and interference with activities of daily living (7 items). Each item was given a score on a numerical scale from 0 (no pain/interference with activities of daily living) to 10 (worst pain imaginable/maximum impact on activities of daily living). The total score for pain intensity is the average of the four pain items. The total score of pain interference is the average score of the seven interference items. The higher score represents high impact.
Time Frame: Month 1
Population: Participants from Prevalence Study Population, participants with the prevalence of breakthrough cancer pain for whom data was collected in prevalence form in the database with breakthrough cancer pain who did not take any treatment for it and who administered the scale. Number analyzed is the participants with data available for the given category.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort 1
Number analyzed (Participants) | 196
score on a scale
  Pain Severity: number analyzed (Participants) | 191
  Pain Severity | 5.33 (1.78)
  Pain Interference: number analyzed (Participants) | 194
  Pain Interference | 6.07 (2.05)

7. Secondary Outcome: Pain Assessment Using the Numeric Rating Scale
Time Frame: Month 1
Population: Data was not collected for this outcome measure.
Arm/Group | Cohort 1
Number analyzed (Participants) | 0

8. Secondary Outcome: Quality of Life Assessment Using the Short Form-12 (SF-12) Questionnaire Score
Description: The SF-12 health questionnaire is a 12 question assessment of functional health and well-being. The survey asks about various health aspects, including physical functioning, role limitations due to physical health problems, bodily pain, general health, vitality, social functioning, role limitations due to emotional problems, and mental health (psychological distress and psychological well-being). Two summary measures are derived: the Physical and the Mental Health Component Summary. For each component summary, survey items were weighted and summed to create a summary score between 0 (poor mental and physical quality of life) and 100 (better mental and physical quality of life).
Time Frame: Month 1
Population: Participants from Prevalence Study Population, participants with the prevalence of breakthrough cancer pain for whom data was collected in prevalence form in the database with breakthrough cancer pain who did not take any treatment for it and who administered the scale with data available for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort 1
Number analyzed (Participants) | 188
score on a scale
  Physical Component SF-12 | 28.53 (7.97)
  Mental Component SF-12 | 36.87 (9.51)

9. Secondary Outcome: Participant's Performance as Assessed by the Karnofsky Scale Score
Description: Karnofsky performance score is used to quantify participant's general well-being and activities of daily life and participants are classified based on their functional impairment. Karnofsky performance score is 11 level score which ranges between 0 (death) to 100 (participant asymptomatic with no evidence of illness). Higher score means higher ability to perform daily tasks. Participants with missing values in the Karnofsky scale were assigned to the worst score of 0, however, in these cases it is not 'death'.
Time Frame: Month 1
Population: Prevalence Study Population included participants with the prevalence of breakthrough cancer pain for whom data was collected in prevalence form in the database with data available for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1
Number analyzed (Participants) | 3751
percentage of participants
  Score 0 | 0.2
  Score 10 | 0.5
  Score 20 | 0.8
  Score 30 | 1.4
  Score 40 | 2.2
  Score 50 | 2.9
  Score 60 | 6.7
  Score 70 | 11.9
  Score 80 | 22.6
  Score 90 | 25.7
  Score 100 | 25.2

ADVERSE EVENTS:
Time Frame: Baseline up to Month 1
Description: Data of adverse events or adverse drug reactions were not collected as part of the study database.
Arm/Group | Cohort 1
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2016-02-19): https://cdn.clinicaltrials.gov/large-docs/84/NCT02899884/Prot_000.pdf
  • Statistical Analysis Plan (2017-01-24): https://cdn.clinicaltrials.gov/large-docs/84/NCT02899884/SAP_001.pdf